CLINICAL TRIAL: NCT04397315
Title: Comparative Evaluation of Partial and Complete Pulpotomy in Mature Permanent Molars With Clinical Signs Indicative of Irreversible Pulpitis
Brief Title: Comparative Evaluation of Partial and Complete Pulpotomy in Permanent Molars
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Dr. Ankita Ramani
Record Dates: First submitted 2020-05-12; First posted 2020-05-21 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Pulpitis - Irreversible
Keywords: Irreversible Pulpitis; Complete Pulpotomy; Partial Pulpotomy; Vital Pulp Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Complete Pulpotomy (Active Comparator): In case of complete pulpotomy procedure the exposed pulp tissue will be amputated using sterile bur in high speed hand piece to the level of canal orifices.
  Interventions: Procedure: Pulpotomy to the level of canal orifices
- Partial Pulpotomy (Active Comparator): In case of partial pulpotomy procedure the exposed pulp tissue will be amputated using a sterile bur in the high speed hand piece to a depth of 2-3 mm.
  Interventions: Procedure: Pulpotomy up to superficial 2-3 mm of pulp chamber

INTERVENTIONS:
Procedure: Pulpotomy to the level of canal orifices — Pulp tissue will be removed till the level of canal orifices.
  Arms: Complete Pulpotomy
Procedure: Pulpotomy up to superficial 2-3 mm of pulp chamber — Only superficial pulp from the chamber will be removed
  Arms: Partial Pulpotomy

SUMMARY:
This study will compare the outcome of partial pulpotomy and complete pulpotomy in mature permanent molars with clinical signs indicative of irreversible pulpitis

DETAILED DESCRIPTION:
After thorough history and clinical and radio graphic examination, and confirmation of eligibility for the study, written informed consent will be taken after explaining the procedure and its associated risks and benefits. Clinical diagnosis of irreversible pulpitis will be established based on a history of spontaneous pain or pain exacerbated by cold stimuli and lasting for a few seconds to several hours (lingering pain) compared to control teeth and which is reproducible using cold testing. Once included, study subjects will be randomly allocated to either Complete Pulpotomy group or Partial Pulpotomy group. (Mineral Trioxide Aggregate) MTA will be used as pulpotomy agent. A layer of resin modified Glass Ionomer liner will be placed over the MTA and tooth will be permanently restored with composite resin in second appointment.

Pain analysis will be carried out preoperatively and postoperatively at every 24 hours till 7 days after intervention. All the subjects will be followed up for evaluation of success at every 3 months from baseline to 1 year.

ELIGIBILITY:
Inclusion Criteria: Inclusion criteria

* The patient should be ≥18 years of age.
* Restorable molar teeth.
* Tooth should give positive response to pulp sensibility testing.
* Clinical diagnosis of irreversible pulpitis.
* Tooth with probing pocket depth and mobility are within normal limits.
* No signs of pulpal necrosis including sinus tract or swelling.
* Non-contributory medical history

Exclusion Criteria:

* Teeth with immature roots.
* No pulp exposure after caries excavation.
* Bleeding could not be controlled in 6 minutes.
* Insufficient bleeding after pulp exposure, the pulp is judged necrotic or partially necrotic.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Clinical Success and radiographic success | Baseline to 12 Months
  CLINICAL SUCCESS CRITERIA:
  Absence of spontaneous pain, discomfort, swelling, sinus tract or tenderness to palpation or percussion.
  RADIOGRAPHIC SUCCESS CRITERIA:
  No pathosis evident on the radiograph such as root resorption, furcal pathosis or new periapical pathosis.
  Periapical Index score 1 or 2 according to Orstavic et al.
  Evaluation of both clinical and radiographic outcome is must for analyzing the actual success of therapeutic technique. Number of participants fulfilling both clinical as well as radiographic success criteria will be considered in success category.

SECONDARY OUTCOMES:
Pain analysis | Baseline to 7 days
  To assess incidence and intensity of pain postoperatively at every 24 hours till 7 days using Visual analogue Scale of 0 to 10 Centimetere line. Score 0 means no pain and Score 10 means maximum pain.

CONTACTS AND LOCATIONS:
Overall Officials: ANKITA RAMANI, Principal Investigator — POST GRADUATE INSTITUTE OF DENTAL SCIENCES, ROHTAK
Locations (1):
- Ankita Ramani, Rohtak, Haryana, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ramani A, Sangwan P. Outcome Following Complete and Partial Pulpotomy in Managing Cariously Exposed Mature Permanent Molars With Symptomatic Irreversible Pulpitis: A 5-Year Follow-Up of a Randomised Clinical Trial. Int Endod J. 2025 Dec;58(12):1835-1848. doi: 10.1111/iej.70028. Epub 2025 Sep 2. PMID 40898413
- [Derived] Ramani A, Sangwan P, Tewari S, Duhan J, Mittal S, Kumar V. Comparative evaluation of complete and partial pulpotomy in mature permanent teeth with symptomatic irreversible pulpitis: A randomized clinical trial. Int Endod J. 2022 May;55(5):430-440. doi: 10.1111/iej.13714. Epub 2022 Mar 10. PMID 35226769